CLINICAL TRIAL: NCT02363010
Title: 1R01DK100345-01A1: An Innovative, Physical Activity-focused Approach to Weight Loss Maintenance
Brief Title: Project Impact: An Innovative Approach to Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Meghan Butryn, Principal Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1402002613
Record Dates: First submitted 2014-09-30; First posted 2015-02-13 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Weight Loss; Overweight
Keywords: Obesity; Weight loss; Overweight
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Behavior Therapy for Weight Loss (Active Comparator): Eighteen months of standard, group-based behavioral treatment for weight loss and weight loss maintenance.
  Interventions: Behavioral: Gold Standard Behavior Therapy for Weight Loss
- Behavior Therapy for Weight Loss with PA emphasis (Experimental): Six months of standard, group-based behavioral treatment for weight loss and weight loss maintenance, followed by 12 months of standard, group-based behavioral treatment for weight loss and weight loss maintenance with a larger emphasis on physical activity goals.
  Interventions: Behavioral: Gold Standard Behavior Therapy for Weight Loss; Behavioral: Behavior Therapy for Weight Loss with Physical Activity Emphasis
- Acceptance-based Behavior Therapy with PA emphasis (Experimental): Six months of standard, group-based behavioral treatment for weight loss and weight loss maintenance, followed by 12 months of group-based behavior therapy with acceptance-based strategies, and a larger emphasis on physical activity goals.
  Interventions: Behavioral: Gold Standard Behavior Therapy for Weight Loss; Behavioral: Acceptance-based Behavior Therapy for Weight Loss with PA emphasis

INTERVENTIONS:
Behavioral: Gold Standard Behavior Therapy for Weight Loss — Group- based behavioral treatment for weight loss and weight loss maintenance, with a standard emphasis on diet (65% of session) and physical activity goals (25% of session). Other weight loss behaviors such as self monitoring will be covered in the remaining time (10% of session).
Behavioral: Behavior Therapy for Weight Loss with Physical Activity Emphasis — Group-based behavioral treatment for weight loss and weight loss maintenance, with a larger emphasis on physical activity goals (65% of session) than eating-related goals (25% of session).Other weight loss behaviors such as self monitoring will be covered in the remaining time (10% of session).
  Arms: Behavior Therapy for Weight Loss with PA emphasis
Behavioral: Acceptance-based Behavior Therapy for Weight Loss with PA emphasis — Group-based, acceptance-based behavioral treatment for weight loss and weight loss maintenance, with a larger emphasis on physical activity goals (65% of session) than eating-related goals (25% of session).Other weight loss behaviors such as self monitoring will be covered in the remaining time (10% of session).
  Arms: Acceptance-based Behavior Therapy with PA emphasis

SUMMARY:
The major goal of this project is to evaluate an innovative approach to obesity. This study will determine if behavioral treatment can be improved by 1) implementing a primary focus on PA following initial weight loss treatment, and 2) using a novel, acceptance-based approach to the promotion of PA.

DETAILED DESCRIPTION:
Most adults who engage in lifestyle modification find it difficult to maintain a high level of PA over the long-term, and most also find that weight regain is inevitable. The current portfolio of available interventions does not adequately address these challenges. This project is designed to test the effectiveness of an intervention that is specifically designed to enhance the ability to maintain, in the long-term, a level of PA high enough to achieve long-term weight loss maintenance.

In the study, 300 obese adults will be recruited from the community and provided with 6 months of group-based, standard behavioral treatment for induction of weight loss (Phase I). A 6-month Phase I was chosen so that all participants will have sufficient time to accomplish initial weight loss before Phase II begins, allowing Phase II to truly be a test of weight loss maintenance. In Phase II, participants will receive one of three interventions, to be delivered for an additional 12 months: 1) behavioral treatment, with the standard emphasis on maintaining changes in diet and PA (BT), 2) behavioral treatment, with a primary emphasis on using these skills to maintain PA (BT-PA), or 3) acceptance-based behavioral treatment, with a primary emphasis on using these skills to maintain PA (ABT-PA).

Assessments will be conducted at baseline, 6 months, 18 months (end of treatment), 24 months (6-month follow-up), and 36 months (18-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI between 27 and 45 kg/m2
* Have the ability to engage in at least 15 minutes of moderate physical activity (e.g. brisk walking)
* Successfully complete all steps in the enrollment process, including attendance at all pre-randomization clinic visits and providing physician clearance

Exclusion Criteria:

* Have a medical condition that prevents safe engagement in moderate-to-vigorous physical activity
* Are lactating, pregnant, or planning to become pregnant in the next three years
* Report recently beginning a course of or changing the dosage of prescription medications that can cause significant weight loss or weight gain
* Are participating in or plan to participate in another weight loss program in the next three years
* Have a primary family member or member of their household participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Butryn, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chabria R, Hagerman CJ, Crane N, Ehmann M, Knudsen FM, Brown KL, Forman E, Butryn ML. Racial disparities in the efficacy of traditional versus acceptance-based behavioral weight loss. Health Psychol. 2025 Jul 24:10.1037/hea0001537. doi: 10.1037/hea0001537. Online ahead of print. PMID 40705619
- [Derived] Butryn ML, Crane NT, Lufburrow E, Hagerman CJ, Forman EM, Zhang F. The Role of Physical Activity in Long-term Weight Loss: 36-month Results From a Randomized Controlled Trial. Ann Behav Med. 2023 Feb 4;57(2):146-154. doi: 10.1093/abm/kaac028. PMID 35640225
- [Derived] Butryn ML, Godfrey KM, Call CC, Forman EM, Zhang F, Volpe SL. Promotion of physical activity during weight loss maintenance: A randomized controlled trial. Health Psychol. 2021 Mar;40(3):178-187. doi: 10.1037/hea0001043. PMID 33630639
- [Derived] Butryn ML, Martinelli MK, Remmert JE, Roberts SR, Zhang F, Forman EM, Manasse SM. Executive Functioning as a Predictor of Weight Loss and Physical Activity Outcomes. Ann Behav Med. 2019 Aug 29;53(10):909-917. doi: 10.1093/abm/kaz001. PMID 30689688
- [Derived] Rosenbaum DL, Clark MH, Convertino AD, Call CC, Forman EM, Butryn ML. Examination of Nutrition Literacy and Quality of Self-monitoring in Behavioral Weight Loss. Ann Behav Med. 2018 Aug 16;52(9):809-816. doi: 10.1093/abm/kax052. PMID 30124757

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Started | 110 | 105 | 105
Completed | 88 | 94 | 89
Not Completed | 22 | 11 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis | Total
Number analyzed (Participants) | 110 | 105 | 105 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 96 | 98 | 289
  >=65 years | 15 | 9 | 7 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.4) | 54.3 (9.01) | 52.7 (10.4) | 52.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 78 | 82 | 250
  Male | 20 | 27 | 23 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 4 | 12
  Not Hispanic or Latino | 107 | 99 | 101 | 307
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 28 | 26 | 26 | 80
  White | 78 | 73 | 73 | 224
  More than one race | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 105 | 105 | 320
BMI [Mean (Standard Deviation); unit: kg/m2] | 35.1 (4.3) | 34.5 (4.6) | 35.8 (5.3) | 35.1 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Objectively measured in the research clinic at each time point on a scale
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: percent weight loss
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 110 | 105 | 105
percent weight loss
  6 Months | 10.5 (5.6) | 10.2 (5.0) | 9.9 (4.7)
  12 Months | 12.3 (8.9) | 12.8 (8.2) | 11.6 (7.8)
  18 months | 10.2 (11.9) | 12.4 (10.1) | 9.1 (10.3)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 12 month weight losses; Test type: Superiority; p = .68, ANOVA — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 18 month weight losses; Test type: Superiority; p = .11, ANOVA — A prior threshold for significance was p<.05; Controlling for baseline weight

2. Primary Outcome: Change in Physical Activity
Description: Objectively measured at each time point using wGT3X-BT accelerometers from Actigraph
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: min per week of MVPA
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 110 | 105 | 105
min per week of MVPA
  Baseline | 64.2 (91.9) | 64.2 (78.6) | 48.6 (73.6)
  6 Months | 133.9 (124.5) | 143.0 (121.0) | 128.8 (115.7)
  12 Months | 129.1 (117.5) | 144.6 (124.9) | 127.3 (126.9)
  18 Months | 110.0 (134.6) | 102.5 (124.0) | 85.9 (101.7)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis; Exploring group differences in 12 month moderator to vigorous physical activity (MVPA); Test type: Superiority; p = .41, Compound Poisson general linear models — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 12 month MVPA; Test type: Superiority; p = .46, Compound Poisson general linear models — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA
Statistical Analysis 3: Comparison: Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 12 month MVPA; Test type: Superiority; p = .82, Compound Poisson general linear models — A priori threshold for statistical significance was p< .05; Controlling for baseline MVPA
Statistical Analysis 4: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis; Exploring group differences in 18 month MVPA; Test type: Superiority; p = .42, Compound Poisson general linear models — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA
Statistical Analysis 5: Comparison: Standard Behavior Therapy for Weight Loss vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 18 month MVPA; Test type: Superiority; p = .28, Compound Poisson general linear models — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA
Statistical Analysis 6: Comparison: Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 18 month MVPA; Test type: Superiority; p = .82, Compound Poisson general linear models — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA

3. Secondary Outcome: Cardiorespiratory Fitness
Description: Time taken to complete a half-mile walk on the treadmill. Shorter times indicate a greater level of cardiorespiratory fitness.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 110 | 105 | 105
sec
  Baseline | 537.1 (98.2) | 576.6 (157.3) | 562.2 (101.8)
  6 months | 503.9 (80.8) | 528.2 (103.7) | 514.1 (73.1)
  12 months | 487.7 (74.7) | 512.2 (96.5) | 500.5 (77.5)
  18 months | 498.0 (80.9) | 518.4 (107.6) | 517.0 (103.7)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 12 month cardiorespiratory fitness, measured by half-mile walk time; Test type: Superiority; p = .06, ANOVA — A priori threshold for statistical significance was p < .05; Controlling for baseline half-mile walk time
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 18 month cardiorespiratory fitness, measured by half-mile walk time; Test type: Superiority; p = .30, ANOVA — A priori threshold for statistical significance was p < .05; Controlling for baseline half-mile walk time

4. Secondary Outcome: Waist Circumference
Description: Measured in the clinical horizontally at the umbilicus.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 110 | 105 | 105
cm
  Baseline | 42.6 (5.5) | 42.6 (4.7) | 41.8 (4.5)
  6 Months | 39.0 (5.1) | 39.7 (4.8) | 38.9 (4.3)
  12 Months | 38.6 (5.2) | 38.8 (4.9) | 38.2 (4.6)
  18 Months | 39.2 (5.8) | 38.9 (5.3) | 38.5 (4.7)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 12 month waist circumference; Test type: Superiority; p = .59, ANOVA — A priori threshold for statistical significance was p < .05; Controlling for baseline waist circumference
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; Exploring group differences in 18 month waist circumference; Test type: Superiority; p = .57, ANOVA — A priori threshold for statistical significance was p < .05; Controlling for baseline waist circumference

5. Other Pre Specified Outcome: Exploratory Moderator: Emotional Overeating
Description: Emotional Overeating Questionnaire. The Emotional Overeating Questionnaire is a six-item self-report questionnaire designed to assess the frequency of emotional overeating (Masheb & Grilo, 2006). Participants rate their frequency of eating an "unusually large amount" over the prior 28 days in response to 6 emotions (anxiety, sadness, loneliness, tiredness, anger, and happiness) on a 7-point Likert scale: 0 = no days, 1 =1-5 days, 2 = 6-12 days, 3 = 13-15 days, 4 = 16-22 days, 5 = 23-27 days, and 6 = every day. Responses to the six items are averaged for a total score. Total scores range from 0-6 (units are scores on the scale). Higher total scores indicate more frequent emotional overeating (i.e., worse outcome). The Emotional Overeating Questionnaire has previously shown high internal consistency (alpha = 0.85) with test-retest reliability among individuals with Binge Eating Disorder (Masheb & Grilo, 2006).
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 103 | 98 | 92
units on a scale
  Baseline | 0.62 (0.83) | 0.58 (0.65) | 0.81 (0.86)
  6 months | 0.50 (0.54) | 0.53 (0.61) | 0.58 (0.60)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Emotional Overeating would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .978, Regression, Linear — A priori threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Emotional Overeating would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .998, Regression, Poison — A priori threshold for statistical significance was p <.05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated
Statistical Analysis 3: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Emotional Overeating would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .878, Regression, Linear — A priori threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 4: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Emotional Overeating would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .602, Regression, Poison — A priori threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated

6. Other Pre Specified Outcome: Exploratory Moderator: Disinhibited Eating.
Description: The 18-item Three Factor Eating Questionnaire (TFEQ) (Cappelleri, Bushmakin, Gerber, Leidy, Sexton, Lowe, et al., 2009) assessed disinhibited eating behavior. The questionnaire consists of statements about food and participants rate if they apply to them on a 4-point Likert scale (definitely true, mostly true, mostly false, definitely false). The questionnaire has a well-validated three-factor structure (Cronbach's α of 0.78-0.94), which includes a domain for disinhibited eating. This project used scoring from Niemeier, Phelan, Fava, & Wing, 2007, responses are coded 0 (mostly/definitely false) or 1 (mostly/definitely true). Total scores range from 0-18 (higher scores mean more problematic eating behaviors, i.e., worse outcome). The disinhibited eating subscale is the sum of 16 items (range 0-16), such as: "Sometimes when I start eating, I just can't seem to stop." Higher scores indicate higher levels of disinhibited eating (i.e., worse outcome). Units are scores on the scale.
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 110 | 101 | 103
units on a scale
  Baseline | 8.50 (3.08) | 8.89 (3.38) | 9.40 (3.61)
  6 months | 7.55 (3.03) | 7.77 (3.27) | 7.54 (3.60)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Disinhibited Eating would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .487, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Disinhibited Eating would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .262, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated
Statistical Analysis 3: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Disinhibited Eating would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .851, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 4: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Disinhibited Eating would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .978, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated

7. Other Pre Specified Outcome: Exploratory Moderator: Hedonic Hunger
Description: The Power of Food Scale is a 15-item self-report questionnaire that assesses the tendency to eat for pleasure (rather than physiological hunger) based on cues from the environment (Lowe et al., 2009). Items measure participants' appetite-related thoughts, feelings, and motivations for highly palatable foods with three subscales based on food proximity: (1) Food available in the environment but not physically present (sum of 6 items, range 6-30) (2) Food physically present but not yet tasted (sum of 4 items, range 4-20), and (3) Food tasted but not yet consumed (sum of 5 items, range 5-25). An example item is: "If I see or smell a food I like, I get a powerful urge to have some." Participants rated each of these statements on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Total scores are a sum of the 15 items (range 15-75) (units are scores on the scale). Higher total and subscale scores indicate greater hedonic hunger (i.e., worse outcome).
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 109 | 101 | 101
units on a scale
  Baseline | 40.00 (13.18) | 38.81 (13.04) | 42.65 (13.83)
  6 months | 39.01 (13.58) | 37.14 (13.11) | 39.04 (12.92)
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Hedonic Hunger would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .796, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Hedonic Hunger would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .481, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated
Statistical Analysis 3: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Hedonic Hunger would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .872, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 4: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = .802, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated

8. Other Pre Specified Outcome: Exploratory Moderator: Appetitive Response to Exercise
Description: Perceived Appetitive Response to Exercise. This was a single item measure, where participants were asked to select which one of these four options best described their experience in the past month: There is no relationship between my level of exercise and my appetite; Exercise helps me control my appetite - I am less hungry when I am exercising regularly; Exercise increases my appetite - I am more hungry when I am exercising regularly; Not applicable because not exercising. This item was constructed by the research team, as no pre-existing measure of this construct was identified. The count and percent of participants within each category (by treatment condition) was calculated. This variable consists of four categorical responses, and thus does not have a minimum/maximum value. None of the response options are considered better or worse than the others. Each option describes separate potential experiences participants may have had in relation to eating/exercise over the past month.
Time Frame: 0 months, 6 months
Population: Number of participants analyzed at 6 months may differ from that at baseline based on differential completion of measures by each participant at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
Number analyzed (Participants) | 93 | 89 | 84
Participants
  Baseline: number analyzed (Participants) | 93 | 84 | 84
  Baseline: Not applicable (I have not exercised). | 16 | 15 | 19
  Baseline: There is no relationship between my level of exercise and my appetite. | 34 | 32 | 34
  Baseline: Exercise helps me control my appetite - I am less hungry when I am exercising regularly. | 26 | 25 | 17
  Baseline: Exercise increases my appetite - I am more hungry when I am exercising regularly. | 17 | 12 | 14
  6 Months: number analyzed (Participants) | 92 | 89 | 84
  6 Months: Not applicable (I have not exercised). | 1 | 3 | 4
  6 Months: There is no relationship between my level of exercise and my appetite. | 35 | 30 | 32
  6 Months: Exercise helps me control my appetite - I am less hungry when I am exercising regularly. | 34 | 37 | 31
  6 Months: Exercise increases my appetite - I am more hungry when I am exercising regularly. | 22 | 19 | 17
Statistical Analysis 1: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Appetitive Response to Exercise would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .926, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 2: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that baseline Appetitive Response to Exercise would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .820, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated
Statistical Analysis 3: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Appetitive Response to Exercise would not significantly moderate the relationship between the three treatment conditions and 36-month weight loss. As a note, multiple imputation for missing weight loss data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .127, Regression, Linear — A prior threshold for statistical significance was p < .05; Controlling for baseline weight
Statistical Analysis 4: Comparison: Standard Behavior Therapy for Weight Loss vs Behavior Therapy for Weight Loss With PA Emphasis vs Acceptance-based Behavior Therapy With PA Emphasis; The null hypothesis was that 6-month Appetitive Response to Exercise would not significantly moderate the relationship between the three treatment conditions and 36-month MVPA. As a note, multiple imputation for missing MVPA data was not conducted for exploratory moderation analyses; Test type: Superiority; p = .814, Regression, Poison — A prior threshold for statistical significance was p < .05; Controlling for baseline MVPA. Poisson linear regression was used as MVPA data distribution was zero-inflated

ADVERSE EVENTS:
Time Frame: 36 months
Description: No serious adverse events occurred.
Arm/Group | Standard Behavior Therapy for Weight Loss | Behavior Therapy for Weight Loss With PA Emphasis | Acceptance-based Behavior Therapy With PA Emphasis
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/110 | 0/105 | 0/105

LIMITATIONS AND CAVEATS:
High attrition; low power to detect small effects; no measurement of dietary intake; imperfect measurements of physical activity; conditions differed on how eating behavior was addressed; underrepresentation of men, racial groups outside of non-Hispanic White or Black, young adults, older adults, and those with low levels of education; conducted as a high-intensity BWL within an academic research clinic which may differ from lower-intensity or community-based formats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02363010/Prot_SAP_000.pdf